CLINICAL TRIAL: NCT03939104
Title: A Multi-centre Randomised Controlled Non-inferiority Trial to Compare the Efficacy, Safety and Tolerability of Triple Artemisinin-based Combination Therapies Versus First-line ACTs + Placebo for the Treatment of Uncomplicated Plasmodium Falciparum Malaria in Asia
Brief Title: A Trial to Compare the Efficacy, Safety and Tolerability of Combinations of 3 Anti-malarial Drugs Against Combinations of 2 Anti-malarial Drugs (Asia)
Acronym: DeTACT-ASIA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Mahidol Oxford Tropical Medicine Research Unit (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MAL18005
Record Dates: First submitted 2019-04-29; First posted 2019-05-06 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2023-05

CONDITIONS: Plasmodium Falciparum Malaria (Uncomplicated)
Keywords: Artemether; Lumefantrine; Amodiaquine; Piperaquine; Artesunate; Mefloquine
MeSH Terms: conditions — Malaria, Falciparum

STUDY DESIGN:
Intervention Model Description: A partially blinded randomised controlled non-inferiority trial comparing the efficacy, tolerability and safety of Triple ACTs artemether-lumefantrine+amodiaquine (AL+AQ) and artesunate- mefloquine+piperaquine (AS-MQ+PPQ) and the ACTs artemether-lumefantrine+placebo (AL+PBO), artesunate-mefloquine+placebo (AS-MQ+PBO) (with single-low dose primaquine in some sites) for the treatment of uncomplicated Plasmodium falciparum malaria to assess and compare their efficacy, safety, tolerability.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Artemether-lumefantrine+amodiaquine (AL+AQ) (Active Comparator): Triple ACTs
  Interventions: Drug: Artemether-lumefantrine+amodiaquine
- Artesunate-mefloquine+piperaquine (AS-MQ+PPQ) (Active Comparator): Triple ACTs
  Interventions: Drug: Artesunate-mefloquine+piperaquine
- artemether-lumefantrine+placebo (AL+PBO) (Active Comparator): ACTs
  Interventions: Drug: Artemether-lumefantrine+placebo
- Artesunate-mefloquine+placebo (AS-MQ+PBO) (Active Comparator): ACTs.
  Interventions: Drug: Artesunate-mefloquine+placebo

INTERVENTIONS:
Drug: Artemether-lumefantrine+amodiaquine — AL: Currently available as dispersible tablets containing 20 mg of artemether and 120 mg of lumefantrine, in a fixed-dose combination formulation. The flavoured dispersible tablet paediatric formulation facilitates use in young children.
  The dose of artemether-lumefantrine is administered approaching the WHO-recommended target ranges of artemether 5-24 mg/kg and lumefantrine 29-144 mg/kg over 3 days.
  AQ: Amodiaquine is available as dispersible tablets of 40 mg. The weight-based treatment schedule aims for a dosage of approximately 10mg (4.5-15mg)/kg/day amodiaquine for three days.
  Arms: Artemether-lumefantrine+amodiaquine (AL+AQ)
Drug: Artemether-lumefantrine+placebo — AL: Currently available as dispersible tablets containing 20 mg of artemether and 120 mg of lumefantrine, in a fixed-dose combination formulation. The flavoured dispersible tablet paediatric formulation facilitates use in young children.
  The dose of artemether-lumefantrine is administered approaching the WHO-recommended target ranges of artemether 5-24 mg/kg and lumefantrine 29-144 mg/kg over 3 days.
  PBO: Placebo tablets for amodiaquine are identical in size, shape and color to the amodiaquine tablets.
  Arms: artemether-lumefantrine+placebo (AL+PBO)
Drug: Artesunate-mefloquine+piperaquine — AS: Artesunate will be administered according to an optimised dosing schedule using tablets of 32 or 100 mg artesunate with a dosing target of 4 mg/kg/day.
  MQ: Mefloquine will be administered according to an optimised dosing schedule using tablets of 70 or 220 mg mefloquine hydrochloride with a dosing target of 8.3 mg/kg/day.
  PPQ: Piperaquine will be administered according to an optimised dosing schedule using tablets of 160 or 500 mg of piperaquine tetraphosphate. The weight-based treatment aims for a dosage of approximately
  * 24 mg/kg/day in patients <25 kg (range 16.0 - 32.0 mg/kg) piperaquine for three days, thereby approaching the WHO-recommended target range of 20 - 32 mg/kg per day.
  * 18 mg/kg/day in patients ≥25 kg (range 15.0 - 29.4 mg/kg) piperaquine for three days, thereby approaching the WHO-recommended target range of 16 - 27 mg/kg per day.
  Arms: Artesunate-mefloquine+piperaquine (AS-MQ+PPQ)
Drug: Artesunate-mefloquine+placebo — AS: Artesunate will be administered according to an optimised dosing schedule using tablets of 32 or 100 mg artesunate with a dosing target of 4 mg/kg/day.
  MQ: Mefloquine will be administered according to an optimised dosing schedule using tablets of 70 or 220 mg mefloquine hydrochloride with a dosing target of 8.3 mg/kg/day.
  PBO: Placebo tablets for piperaquine are identical in size, shape and colour to the piperaquine tablets.
  Arms: Artesunate-mefloquine+placebo (AS-MQ+PBO)

SUMMARY:
A partially blinded randomised controlled non-inferiority trial comparing the efficacy, tolerability and safety of Triple ACTs artemether-lumefantrine + amodiaquine (AL+AQ) and artesunate- mefloquine+piperaquine (AS-MQ+PPQ) with the ACTs artemether-lumefantrine + placebo (AL+PBO) and artesunate- mefloquine + placebo (AS-MQ+PBO) (with single-low dose primaquine in some sites) for the treatment of uncomplicated Plasmodium falciparum malaria to assess and compare their efficacy, safety, tolerability.

DETAILED DESCRIPTION:
Subjects will be randomized to up to four arms: artemether-lumefantrine + amodiaquine, artemether-lumefantrine + placebo, artesunate-mefloquine + piperaquine and artesunate-mefloquine + placebo. As a contingency measure in case of significant differences in the efficacy or safety of one of the combinations being tested and/or study drug expiry or unavailability, subjects may be randomised to 2 arms with a matching ACT-TACT pair, i.e., with artemether-lumefantrine + placebo or artemether-lumefantrine + amodiaquine OR artesunate-mefloquine + placebo or artesunate-mefloquine + piperaquine.

Some sites may randomize between 2 arms only with matching ACT-TACT pairs, i.e., artemether-lumefantrine + placebo or artemether-lumefantrine + amodiaquine OR artesunate-mefloquine + placebo or artesunate-mefloquine + piperaquine.

In the control arms, the ACT will be co-packed with a matched (appearance) placebo.

In lower transmission settings (Annual Parasite Incidence <50 per 1000 population per year) the treatment will include a single 0.25 mg/kg gametocytocidal dose of primaquine as recommended by the WHO for children ≥10 kg. All drug administrations will be observed.

Subjects will be treated in an in-patient unit for 3 days and followed up weekly up to D63. Microscopy to detect and quantify malaria parasitaemia will be performed daily (more frequently in patients with parasite density of >5000/µL at inclusion) during hospitalization, at all weekly and unscheduled visits. A physical examination and measurements of vital signs along with a symptom questionnaire for tolerability will be performed and recorded through a standardized method at baseline, daily during admission and weekly during follow up through D42 and at all unscheduled visits. Physical exam, vital sign measurements and assessments of symptoms will be performed on D49, D56, and D63 only for patients who are parasitaemic or those who report fever or other symptoms. Electrocardiographs will be performed during admission (H0, H4, H52, or H64) and day 42 of follow up to assess and compare the effect of ACTs and TACTs antimalarials on QT or QTc-intervals.

The DeTACT-ASIA Trial is funded by UK Aid from the UK government's Foreign, Commonwealth and Development Office (FCDO). The FCDO project number is 300341-114.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, >/= 6 months
* Ability to take oral medication
* Acute uncomplicated P. falciparum monoinfection
* Asexual P. falciparum parasitaemia: 96 to 200,000/µL, determined on a peripheral blood film
* Fever defined as >/= 37.5°C tympanic temperature or a history of fever within the last 24 hours
* Written informed consent by the subject or parent/guardian in case of children lower than the age of consent and assent if required (per local regulations)
* Willingness and ability of the subjects or parents/guardians to comply with the study protocol for the duration of the study

Exclusion Criteria:

* Signs of severe malaria (adapted from WHO criteria)
* Patients not fulfilling criteria for severe malaria but with another indication for parenteral antimalarial treatment at the discretion of the treating physician
* Haematocrit < 20% at screening
* Subjects who have received artemisinin or a derivative within the previous 7 days OR lumefantrine or amodiaquine within the previous 14 days OR mefloquine or piperaquine within the previous 30 days
* Acute illness other than malaria requiring systemic treatment
* Severe acute malnutrition
* Known HIV infection
* Known tuberculosis infection
* For females: pregnant, trying to get pregnant or are lactating
* History of allergy or known contraindication to any of the study drugs, including neuropsychiatric disorders and epilepsy
* Previous splenectomy
* Enrolment in DeTACT in the previous 3 months
* Participation in another interventional study in the previous 3 months

Criteria for severe malaria

* Impaired consciousness (Glasgow Coma Scale, Blantyre Coma Scale)
* Prostration
* Respiratory distress (defined as maximal respiratory rate, by age)
* ≥2 convulsions in the past 24 hours
* Circulatory collapse
* Pulmonary edema
* Abnormal bleeding
* Visible jaundice
* Haemoglobinuria (blackwater)
* Hyperparasitaemia (>10%)

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2023-01-06 (Actual); Study Completion 2023-01-28 (Actual)

PRIMARY OUTCOMES:
Efficacy defined as PCR corrected adequate clinical and parasitological response (ACPR). | 42 days

SECONDARY OUTCOMES:
Efficacy defined as PCR corrected adequate clinical and parasitological response (ACPR) | 63-day
Efficacy defined as adequate clinical and parasitological response (PCR) | 63-day
Efficacy defined as adequate clinical and parasitological response (ACPR) | 42-day
Parasite clearance half-life | 7 days
proportion of subjects with microscopically detectable P. falciparum parasitaemia | 3 days
Fever clearance time | 7 days
  Time taken for the tympanic temperature to fall below 37.5 ºC in patients who were febrile at inclusion
Proportion of subjects with gametocytemia during and after treatment stratified by presence of gametocytes at enrolment | 63 days
Number of adverse events | 42 days
Number of serious adverse events | 42 days
  Including markers of hepatic, renal or bone marrow toxicity
Number of cardiotoxicity events | 52 or 64 hours depends on treatment arm
  In particular QTc-interval above 500 ms or an increase > 60 ms above baseline values at timepoint H4 and H52/H64 and between these time points
Change in haemoglobin stratified for G6PD status/genotype | 28 days
Proportion of subjects requiring retreatment due to vomiting within 1 hour after administration of the study drugs | 1 hour
Proportion of subjects that reports completing a full course of observed TACT | 3 days
Proportion of subjects that reports completing a full course of observed ACT | 3 days
Pharmacokinetic profiles and interactions (including Cmax) of artemisinin-derivatives and partner drugs in ACT and TACT treated subjects in correlation with pharmacodynamics measures of drug efficacy | 42 days
Pharmacokinetic profiles and interactions (AUC) of artemisinin-derivatives and partner drugs in ACT and TACT treated subjects in correlation with pharmacodynamics measures of drug efficacy | 42 days
Plasma levels of partner drugs in correlation with treatment efficacy and treatment arm | 7 days

OTHER OUTCOMES:
Comparison of efficacy, defined as PCR corrected adequate clinical and parasitological response (ACPR) at day 42 versus day 63 | 63 days
Comparison of efficacy, defined as adequate clinical and parasitological response (ACPR) at day 42 versus day 63 | 63 days
Proportions of recurrent infections with parasites carrying mutations of known functional significance | 63 days
Proportions of specimens collected at baseline with parasites carrying mutations of known functional or operational significance | baseline
  Mutations include pfkelch13, pfcrt, pfmdr1, pfdhfr, pfdhps, pfplasmepsin2 , partial or complete deletions of pfhrp2 and other current parasite genetic markers associated with resistance or identified over the course of the study
Number of samples from drug sensitive and resistant parasites that have common genomic patterns that associate with in vivo or in vitro parasite drug sensitivity phenotypes. | 63 days
Survival rate or IC50 in in vitro drug susceptibility assay of P. falciparum to artemisinins and partner drugs according to study sites and genotype | 63 days
Percent agreement and/or KAPPA score of SNPs assessed from dry blood spots versus from whole genome sequencing in leukocyte depleted blood samples | 63 days
Correlation between qPCR based versus microscopy based assessments of parasite clearance dynamics | 14 days
Correlation of parasite clearance metrics as assessed by microscopy versus digital microscopy | 3 days
Number of samples from drug sensitive and resistant parasites obtained before treatment and 6, 12, and 24 hours after start of treatment that can be assigned to a common transcriptomic pattern. | 63 days
Levels of RNA transcription coding for male or female specific gametocytes at admission up to day 14, stratified by the presence of gametocytes at enrolment | 14 days
Correlation between the host genotype and the pharmacokinetics and pharmacodynamics of antimalarials | 42 days
  Host genotype (e.g., CYP2D6, CYP3A4, KCNQ1/LQT1, KCNH2/LQT2, SCN5A/LQT3)
Correlations between the place of residence, work, recent travel history assessed by interview and mobile phone records to identify behaviours and risk factors associated with malaria infection. | 63 days
Correlation between titres of antibodies against malaria parasite antigen and efficacy defined as PCR corrected adequate clinical and parasitological response (ACPR) | 63 days
Correlation between titres of antibodies against malaria parasite antigen and efficacy defined as adequate clinical and parasitological response (ACPR) | 63 days

CONTACTS AND LOCATIONS:
Locations (3):
- Ramu Upazilla Health Complex, Cox’s Bāzār, Chittagong, Bangladesh
- Cambodia (2):
  - Kravanh Referral Hospital, Phnum Kravanh, Pursat
  - Siem Pang Health Center, Siem Pang, Stung Treng

IPD SHARING:
Plan to Share IPD: Yes
With participant's consent, participant's data and results from blood analyses stored in the database may be shared according to the terms defined in the MORU data sharing policy with data repositories such as the WorldWide Antimalarial Resistance Network (WWARN, terms of submission here: http://www.wwarn.org/tools-resources/terms-submission) or other researchers to use in the future. All personal information will be anonymised so that no individual can be identified from their treatment records, through interviews, or from mapping data.
Time Frame: After completion of trial activities and reporting
Access Criteria: MORU Data Sharing Policy: https://www.tropmedres.ac/units/moru-bangkok/bioethics-engagement/data-sharing WWARN terms of Data Access: http://www.wwarn.org/tools-resources/terms-reshouces/terms-data-access
URL: https://www.tropmedres.ac/units/moru-bangkok/bioethics-engagement/data-sharing/moru-tropical-network-policy-on-sharing-data-and-other-outputs

DOCUMENTS (2):
  • Study Protocol (2022-03-23): https://cdn.clinicaltrials.gov/large-docs/04/NCT03939104/Prot_001.pdf
  • Statistical Analysis Plan (2024-03-11): https://cdn.clinicaltrials.gov/large-docs/04/NCT03939104/SAP_002.pdf